CLINICAL TRIAL: NCT05460520
Title: Developing Robust Treatment Options for Mal de Débarquement Syndrome
Brief Title: DevRobust Treatment for Mal de Débarquement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: New York University (Other); Brooklyn College of the City University of New York (Other); Ohio University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Sergei Yakushin, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 21-0162; R01DC019928 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mal de Débarquement Syndrome

STUDY DESIGN:
Intervention Model Description: Qualified applicants with dominant oscillatory motion sensations will be randomly assigned to Groups 1 (n=50), 2 (n=50), 3 (n=30), or 4 (n=30), and those with dominant gravitational pull sensation will be randomly assigned to groups 5 (n=20) or 6 (n=20).
Who Masked: Participant, Outcomes Assessor
Masking Description: The group assignment will be based on a random drawing of numbers prepared by Dr. Maruta, to the outcome of which he will be blinded. Dr. Cho (NYU) will interview each participant over the phone prior and at the completion of the final 6-month follow-up to independently record symptom severity scores as reported by the participants. Dr. Cho will be blinded to the type of the treatment that the participants received. Dr. Maruta will perform analyses of objective (posture, rotational test, VNG) and subjective (DHI, SVQ, VVAS, HADS, STAI etc.) data obtained during the treatment and at follow-ups. Dr. Maruta will be blinded to the participants' identity and the type of treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: VOR readaptation with full-field OKS (Sham Comparator): This group to undergo VOR readaptation with full-field OKS. Groups 1 will be treated with stationary OKS (sham). (Group 1, n=50).
  Interventions: Behavioral: VOR Readaptation
- Group 2: VOR readaptation with VR googles (Sham Comparator): This group to undergo VOR readaptation with VR googles. Groups 2 will be treated with stationary OKS (sham). (Group 2, n=50)
  Interventions: Behavioral: VOR Habituation
- Group 3: Supplemental VOR habituation (Active Comparator): This group to undergo VOR readaptation with full-field OKS combined with a habituation protocol. (Group 3, n=30)
  Interventions: Behavioral: VOR Readaptation; Behavioral: VOR Habituation
- Group 4: Visual desensitization treatment (Active Comparator): This group to undergo VOR readaptation with full-field OKS combined with visual desensitization protocol. (Group 4, n=30)
  Interventions: Behavioral: VOR Readaptation; Behavioral: Visual Motion Desensitization
- Group 5: Treatment of gravitational pull with OKS with full-field setting (Active Comparator): This group with phantom sensation dominated by gravity pull. This group will undergo OKS in a full-field (Group 5, n=20) .
  Interventions: Behavioral: Opposing visual motion stimulus
- Group 6: Treatment of gravitational pull with OKS with VR setting (Active Comparator): This group with phantom sensation dominated by gravity pull. This group will undergo OKS in a VR setting (Group 6, n=20).
  Interventions: Behavioral: Opposing visual motion stimulus

INTERVENTIONS:
Behavioral: VOR Readaptation — The stimulus will be a combination of horizontal visual motion and a head maneuver. The subject will sit in a stationary chair, and a treatment provider will stand behind the subject. While the subject views the slow horizontal motion up to 10°/s of vertical stripes, the provider will gently hold the head of the subject above the ears and tilt the head in the roll (side-to-side) or pitch (up-down) plane by approximately ±20° at the frequency of 0.2 to 0.05 Hz for up to 10 min. The treatment will be repeated with breaks of approximately 5 min. A treatment session will last no longer 120 min including the breaks.
  In Groups 1, 3, and 4, subjects will sit in a chair placed in the center of a cylindrical enclosure of a 95 cm radius, and full-field visual motion will be generated with light projected on the wall of this chamber. In Group 2, visual motion will be presented on the screen of a VR headset. Unlike groups 3 and 4, groups 1 and 2 do not receive any complementary treatment.
  Arms: Group 1: VOR readaptation with full-field OKS; Group 3: Supplemental VOR habituation; Group 4: Visual desensitization treatment
Behavioral: VOR Habituation — The subject will sit in a chair placed in the center of a cylindrical enclosure of a 95 cm radius. Physical motion will be generated by rotating the chair sinusoidally to the left and right, and full-field visual motion will be generated with light projected on the wall of this chamber. Velocity storage will be weakened by inducing a conflict between physical and visual motions. Subjects will be first treated with a stimulus with a peak speed of 5°/s. The stimulus speed will be gradually increased from 5°/s on Day 1 to 40°/s on Day 5. In total, the subjects are expected to undergo 200-280 min of treatment over the five days, broken up into several 10-20 min sessions per day with a 10-min break in between. If signs or symptoms of motion sickness are reported by the subject (nausea, sweating), the session will be immediately paused. Treatment may be continued after a short rest if the discomfort is alleviated or on the following day.
  Arms: Group 2: VOR readaptation with VR googles; Group 3: Supplemental VOR habituation
Behavioral: Visual Motion Desensitization — The subject will be situated in darkness and view the movement of a visual pattern presented on a disk, sized 1 m in diameter and placed 1 m away from the subject with its center at the eye level. The disk will be rotated clockwise and counter-clockwise for up to 10 min at a fixed maximal speed within a treatment session but varying across sessions between 5 to 60°/s. Within a single session, the visual stimulus will be first presented with the subject sitting upright in a chair, and then the treatment will be repeated with the subject standing. The disk will be mounted on a vertical sled, so the center of rotation can be kept at the eye level when sitting and standing. A treatment session will be repeated or conducted with an increased visual motion speed up to 60°/s according to the subject's readiness. In total, the subjects are expected to undergo up to 300 min of treatment over the five days, broken up into several sessions per day with a 10-min break in between
  Arms: Group 4: Visual desensitization treatment
Behavioral: Opposing visual motion stimulus — The investigators characterize gravitational pull as a misaligned sense of upright in the velocity storage mechanism, and hypothesize that that this misalignment can be corrected with an opposing visual motion stimulus, e.g., backward pulling will be corrected with upward visual motion.
  Patients in Group 5 will undergo view visual motion in a physical setting, and those in Group 6 under a VR setting. In total, the subjects are expected to undergo up to 300 min of treatment over the five days, broken up into several sessions of 1-10 min per day with an approximately 5-min break in between.
  Arms: Group 5: Treatment of gravitational pull with OKS with full-field setting; Group 6: Treatment of gravitational pull with OKS with VR setting

SUMMARY:
Mal de Débarquement Syndrome (MdDS) is an under-recognized balance disorder, which is manifested by persistent false sensations of oscillatory self-motion (rocking/swaying) and/or pulling in a specific direction (gravitational pull). Patients with MdDS typically experience additional presumably secondary symptoms, such as heightened sensitivity to visual motion (visually induced dizziness, VID), physical motion (motion sickness, MS), and other debilitating physical, cognitive, or affective problems. MdDS was previously considered intractable, and only recently was a breakthrough made in the clinical laboratory with an introduction of a visual-vestibular therapy protocol, yielding a significant long-term improvement of symptoms, including complete remission, in about 50% of patients. However, the approach is limited in several ways. Firstly, there is a practical limitation in implementing the treatment protocol, which requires a specialized set-up for visual stimulation in a dedicated room. This research will address this limitation by testing the utility of virtual reality technology to implement the treatment protocol. Secondly, patients often retain residual symptoms of VID and MS susceptibility, which often act as a trigger for the recurrence of MdDS. This limitation will be addressed by supplementing the original approach with an additional treatment focusing on VID or MS susceptibility. Thirdly, although the original protocol focused on reducing rocking/swaying sensations, gravitational pull often co-occurs with such sensations, and some experience only that motion sensation. This limitation will be addressed by modifying the original protocol. Two hundred patients with MdDS will be recruited for the study. Bias will be controlled by randomized group assignment and the use of placebo treatments. Patients will be treated for 1-2 hours a day for 5 days. Patients will be followed for up to 6 months. The proposed study will facilitate improved outcomes for MdDS by broadening its treatment options.

DETAILED DESCRIPTION:
Objectives This study aims to improve outcomes of MdDS by broadening its treatment options. Specifically, to improve access to the VOR readaptation treatment, the investigators will test the efficacy of VR goggles in generating visual motion to treat MdDS. If proven to be effective, MdDS patients can be treated locally in many vestibular therapy offices, not only for initial treatment but also for remedial or follow-up treatment when symptoms return. To improve long-term outcomes of MdDS, the investigators will evaluate the efficacy of the treatment of a complementary approach combined with VOR readaptation. The investigators hypothesize that an additional intervention that reduces (habituates) the velocity storage capacity will decrease sensitivity to physical movement and improves MdDS symptoms as well as limits symptom recurrence. In addition the investigators hypothesize that desensitization to visual stimuli can reduce visually induced dizziness frequently observed in patients with MdDS. The investigators will verify whether these complementary treatments will provide a better outcome compared to the readaptation treatment by itself. Lastly, to broaden the scope of the VOR readaptation treatment, the study will address the false sensation of gravitational pull commonly reported by patients. The investigators also hypothesize that a visual motion stimulus without cross-axis head motion can reduce this sensation.

Specific Aims Specific Aim 1: Evaluate the efficacy of VR goggles for VOR readaptation. One hundred patients with oscillatory self-motion sensations will be randomly assigned to undergo VOR readaptation with full-field OKS (Group 1, n=50) or VR goggles (Group 2, n=50). Immediate and up to six-month follow-up results will be compared.

Specific Aim 2: Evaluate the efficacy of habituation and visual desensitization combined with VOR readaptation. Sixty patients with oscillatory self-motion sensations will be randomly assigned to undergo VOR readaptation with full-field OKS combined with a habituation (Group 3, n=30) or visual desensitization (Group 4, n=30) protocol. Immediate and up to six-month follow-up results will be compared to those of Group 1.

Specific Aim 3: Treatment of gravitational pull sensation. The investigators estimate that 40 of 200 patients screened for this study will have a phantom sensation dominated by gravity pull, 20 with only that sensation. These patients will be randomly assigned to undergo OKS in a full-field (Group 5, n=20) or VR setting (Group 6, n=20). Immediate and up to six-month follow-up results will be compared.

How Research Will Be Introduced to Participants:

The study will be introduced to potential participants through public announcements such as ClinicalTrials.gov, referrals from clinicians, or direct contact by investigators to individuals who previously requested to be contacted for the opportunity to participate in an MdDS treatment study.

How Participants Will Be Screened:

Informed consent form will be emailed to individuals interested in study participation. Individuals will be contacted by the investigators over the phone and consented for study participation. Consented potential participants will receive intake forms via email with questions regarding the history and symptom characteristics of MdDS, age, sex, and general medical history. Investigators will review the returned intake forms to determine eligibility for study participation based on the inclusion/exclusion criteria described separately and a telephone interview for confirmation and clarification of the candidate's MdDS symptoms. A nystagmography test will then be requested to verify normal inner ear and central vestibular functioning. When candidates do not qualify for the study, screening data will be de-identified, and only those about MdDS symptom presentation, age, sex, and the reason for exclusion will be kept. Intake form and the nystagmography report of the candidates will be securely transferred to NYU for Dr. Catherine Cho to review. Dr. Cho will then conduct a telephone interview with each candidate, and provide PI with confirmation or denial of candidate eligibility, after which the information reviewed by Dr. Cho will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Conformable diagnosis of Mal de Débarquement Syndrome including significant improvement of symptoms with passive motion.

Exclusion Criteria:

* A history of abnormal inner ear or central vestibular function indicated by abnormal nystagmography test (abnormal saccades or pursuit, VOR suppression index <85%, no caloric response, decay time constant of response to rotation less than 10 seconds, spontaneous nystagmus).
* Confounding neurological disorders (e.g., multiple sclerosis, Parkinson's, epilepsy, blindness etc.).
* A history of leg, spine, or other injuries that affect their ability to stand or walk without assisting support.
* High level of anxiety as indicated by State-Trait Anxiety Inventory (≥75) and the Beck Anxiety Inventory (≥55).
* Claustrophobia.
* Patients previously treated with VOR readaptation technique are excluded.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective severity of MdDS-related Symptoms Self-score | Baseline and 6 months
  The levels of subjective severity of MdDS-related symptoms will be reported on an 11-point Likert scale of 0-10, where 0 is no symptoms, and 10 is the most challenging sensation of that symptom that the patient can imagine. Higher score indicates poorer health outcome.

SECONDARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) | Baseline and 6 months
  The form contains 25 questions subdivides into 3 groups to determine the physical, emotional, and functional aspects of disability related to MdDS. Total score range 0-100. Sub-scores: physical disability: 0-24; emotional disability: 0-36; functional disability 0-40. Higher score indicates poorer/better health outcome.
Change in Visual Vertigo Analogue Scale (VVAS) | Baseline and 6 months
  The form contains 9 questions scored 0-10 related to VID. Scores are averaged across all questions. Score >3 - low VID; 3-8 - high VID; >8 - extreme VID. Higher score indicates poorer health outcome.
Change in Situational Vertigo Questionnaire (SVQ) | Baseline and 6 months
  The form Contain 19 questions (scored 0-4) to determine sensitivity to physical motion. Individual scores are averaged. Score <1- not sensitive; 1-3 - sensitive to motion; >3 - highly sensitive to motion. Higher score indicates higher sensitivity to motion.
Change in Beck Anxiety Inventory (BAI) | Baseline and 6 months
  The form contains 21 questions related to anxiety. Each question is ranged 0-3. Individual scores are summated. Total score 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety. Higher score indicates poorer health outcome.
Postural stability | During 5 days of treatment
  Static posturography will be obtained with a custom-designed computer program for a Wii board (Nintendo). The displacement of the center of pressure (COP) over a 1 min period will be measured, and the root means square (RMS) of the postural displacement will be computed to compare the postural stability before and after the treatment. The total trajectory length (maximum excursion) of the COP deviation over 20 s will also be computed. Postural stability will be measured with the subject standing with their feet 30 cm apart and eyes either open or closed.
Velocity storage time constant | During 5 days of treatment
  The time constant (Tc) of velocity storage will be determined from the decay profile of the nystagmus's slow phase velocity generated in response to a rotational step velocity of 60°/s in clockwise and counterclockwise directions in darkness. Movements of the right eye will be recorded with video oculography at a rate of 60 frames/s (ISCAN) or binocularly at 250 fr/s (FNND Inc). After 60 s of rotation, the chair will be stopped, and post-rotatory nystagmus will be recorded to 60 s. The total duration of the test is 5 min. The test will be performed before and after daily habituation sessions.
Anonymous REDCap survey | At 6-month follow-up
  Survey contains information on group and whether treatment was effective initially and 6-months after: 1) strongly agree; 2) somewhat agree; 3) cannot determine difference; 4) symptoms slightly worsened; 5) significantly worsened.
Change in the State-Trait Anxiety Inventory (STAI) | Baseline and 6 months
  A 40 self-report items questionnaire, each item scored on 4-point likert-type response scale from 1 (not at all) to 4 (almost always), full range from 20 to 80, with higher score STAI scores suggesting higher levels of anxiety.
Change in The Hospital Anxiety and Depression Scale (HADS) | Baseline and 6 months
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item, 4-point scale to assess depression and anxiety based on the total score of 7 items each. Each item is scored 0 - 3, with full range from 0 to 42, with higher score indicating more severe anxiety or depression.
Change in The Vestibular Disorders Activities of Daily Living Scale (VADL) | Baseline and 6 months
  The Vestibular Disorders Activities of Daily Living Scale (VADL) is a 31-item, 10-point scale to assess functional limitation or disability in people with vestibular disorders focused on essential functional skills and important mobility and instrumental skills. Full score from 1-10, with higher score indicating poorer health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Yakushin, PhD, Principal Investigator — Ichan Scool of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Proposals should be directed to sergei.yakushin@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years at a third party website (tbd).

REFERENCES:
- [Background] Yakushin SB, Raphan T, Cho C. Treatment of Gravitational Pulling Sensation in Patients With Mal de Debarquement Syndrome (MdDS): A Model-Based Approach. Front Integr Neurosci. 2022 May 23;16:801817. doi: 10.3389/fnint.2022.801817. eCollection 2022. PMID 35676926
- [Background] Yakushin SB, Zink R, Clark BC, Liu C. Readaptation Treatment of Mal de Debarquement Syndrome With a Virtual Reality App: A Pilot Study. Front Neurol. 2020 Aug 18;11:814. doi: 10.3389/fneur.2020.00814. eCollection 2020. PMID 33013617
- [Background] Dai M, Cohen B, Cho C, Shin S, Yakushin SB. Treatment of the Mal de Debarquement Syndrome: A 1-Year Follow-up. Front Neurol. 2017 May 5;8:175. doi: 10.3389/fneur.2017.00175. eCollection 2017. PMID 28529496